CLINICAL TRIAL: NCT03236506
Title: A Direct obserVed therApy vs fortNightly CollEction Study for HCV Treatment - ADVANCE HCV Study
Acronym: ADVANCE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Dundee (Other)
Responsible Party: Principal Investigator, John Dillon, Professor John Dillon, University of Dundee
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016GA03; 2017-001039-38 (EudraCT Number)
Record Dates: First submitted 2017-07-04; First posted 2017-08-02 (Actual); Results first posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-10

CONDITIONS: Hepatitis C
Keywords: Illicit drug; Injecting drug
MeSH Terms: conditions — Hepatitis C; Substance-Related Disorders | interventions — elbasvir; grazoprevir; elbasvir-grazoprevir drug combination; Psychosocial Intervention; Sofosbuvir

STUDY DESIGN:
Intervention Model Description: Randomised, un-blinded trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Daily observed therapy (Experimental): Patients with active hepatitis C infection genotype 1 will receive 12 weeks treatment with Zepatier at one tablet per day. Patients with active hepatitis C infection genotype 3 will receive 8 weeks treatment with Zepatier pill plus Sofosbuvir pill at one of each tablets per day. These tablets will be given to patients on a daily, observed basis by either the nurse or a community pharmacist.
  Interventions: Drug: Elbasvir/Grazoprevir 50 MG-100 MG Oral Tablet; Drug: Sofosbuvir 400 MG
- Fortnightly pick-up (Active Comparator): Patients with active hepatitis C infection genotype 1 will receive 12 weeks treatment with Zepatier at one tablet per day. Patients with active hepatitis C infection genotype 3 will receive 8 weeks treatment with Zepatier pill plus Sofosbuvir pill at one of each tablets per day. These tablets will be given to patients on a fortnightly basis by the nurse.
  Interventions: Drug: Elbasvir/Grazoprevir 50 MG-100 MG Oral Tablet; Drug: Sofosbuvir 400 MG
- Fortnightly pick-up +psych intervention (Active Comparator): Patients with active hepatitis C infection genotype 1 will receive 12 weeks treatment with Zepatier at one tablet per day. Patients with active hepatitis C infection genotype 3 will receive 8 weeks treatment with Zepatier pill plus Sofosbuvir pill at one of each tablets per day. These tablets will be given to patients on a fortnightly basis by the nurse. In addition, this group will receive a one-off interview with the researcher to complete a psychological intervention designed to improve adherence to the medication regimen.
  Interventions: Drug: Elbasvir/Grazoprevir 50 MG-100 MG Oral Tablet; Behavioral: Psychological intervention; Drug: Sofosbuvir 400 MG

INTERVENTIONS:
Drug: Elbasvir/Grazoprevir 50 MG-100 MG Oral Tablet — Drugs will be given to participants to treat hepatitis C infection
  Other Names: Zepatier
Behavioral: Psychological intervention — Participants randomised to fortnightly pick-up with psychological intervention will have an interview with the study nurse designed to aid their compliance with the drug regimen. During the intervention participants will be guided by their trial nurse in the completion of a personalised booklet, "Hepatitis C and Me". The booklet uses the principles of node-link mapping to structure the intervention.
  Arms: Fortnightly pick-up +psych intervention
Drug: Sofosbuvir 400 MG — Drugs will be given along with Zepatier to participants to treat genotype 3hepatitis C infection
  Other Names: Sovaldi

SUMMARY:
Hepatitis C is a blood borne virus that can seriously damage the liver. An estimated 50,000 Scots have been infected with Hepatitis C virus (HCV). The main driver for spread of HCV infection is intravenous drug use. As HCV is highly infectious by the blood borne route through needle sharing, it can infect the person who injects drugs (PWID) early in their habit.

Around two thirds of people who are infected are unaware of it, and often show no symptoms over a long period of time. While there is presently no vaccination for Hepatitis C, improved treatments with shorter duration are now available. This raises the possibility of using therapy as prevention, turning the epidemic off at source, by targeting active PWID who are the main source of new infections. Modelling work illustrates the startling possibility and impact of treating drug users to reduce the prevalence of HCV.

The focus of this trial will be to ascertain whether oral treatment regimens are effective in the treatment as prevention scenario in an active PWID population where illicit drug taking and poor adherence may reduce treatment efficacy. The investigators will trial 3 different methods of delivering treatment and will trial an unlicensed combined treatment against HCV genotype 3 infection of shortened duration since current regimens for this genotype are limited.

The investigators will recruit 135 participants and randomise them to one of three arms: daily, directly observed therapy; fortnightly dispensing of drugs; fortnightly dispensing of drugs with a psychological adherence intervention. Randomisation will be stratified according to HCV genotype. Participants will be treated for 12 or 8 weeks depending on genotype and followed up 12 weeks post treatment for the measurement of sustained viral response (SVR). The primary outcome measure will be SVR at 12 weeks post treatment (SVR12), as this measure of cure is the determinant of sufficient compliance and efficacy within the 3 treatment arms. Analysis will be by modified intention to treat of all participants who receive one dose of therapy, to show non-inferiority fortnightly dispensing is easier to deliver than daily dispensing.

DETAILED DESCRIPTION:
Hepatitis C is a blood borne virus that can seriously damage the liver. An estimated 50,000 Scots have been infected with Hepatitis C virus (HCV). The main driver for spread of HCV infection is intravenous drug use. As HCV is highly infectious by the blood borne route through needle sharing, it can infect the PWID early in their habit. With the advent of more effective therapies of shortening duration, it raises the possibility of using therapy as prevention, turning the epidemic off at source, by targeting active infected drug users who are the main source of new infections.

The modelling work of Martin et al, raises the startling possibility of the profound impact of treating small numbers of drug users on the prevalence of HCV, the work shows that treating as few as 10-20 per 1000 drug users per year can reduce HCV prevalence by 50-90% over 10 years. This has generated in the HCV field, the concept of treatment as prevention. The scale of the benefit is exponentially related to prevalence of HCV in the population, the lower the prevalence the bigger the impact. The model has some limitations, it groups all drug users together and assumes a similar risk of infection for those on methadone and those actively injecting and assumes a high rate of turn over from methadone back to active injecting and further assumes treatment is only possible during the opiate substitution phase.

Oral anti-HCV regimens that are interferon free and have virtually no side-effects are now the standard of care in conventional treatment populations. The medication should be taken daily to optimise therapeutic success, and if adherence is poor in the actively injecting population it is possible that the effectiveness of the new oral drugs will be reduced. It is key to know if all oral directly acting antivirals (DAA) regimens are robust and maintain SVR rates in this population. The real world SVR rate combined with drug cost, re-infection rate and emergence of viral resistance will determine if this treatment as prevention model is cost-effective with DAAs. Directly observed therapy (DOT) is the ultimate adherence aid, but it is more costly and draconian so that it may discourage participants, especially this group, from taking up therapy. Therefore the investigators need to demonstrate that treatment uptake and adherence is sufficient to maintain the SVR rate at a level which makes treatment as prevention cost effective. Three means of delivery will be compared: daily DOT vs fortnightly pick up of therapy vs. fortnightly pick-up of therapy with a psychological intervention for adherence. The DOT method of treatment has not been explored in this difficult to find and engage population previously. Contingency management in the form of protein drinks for successful completion of each fortnight of treatment will be provided in all three arms of the trial. A comparison of the three pathways mentioned above will show which pathway shows best acceptability to participants and greatest compliance

The advent of DAAs with their reduced side effect profiles, shorter treatment duration and high SVR rates have the potential to reduce the burden of treatment providing high levels of adherence can be maintained. However, the use of DAAs alone are unlikely to be sufficient to achieve the required levels of adherence. In addition, the use of DAAs will not address the psychosocial factors known to influence adherence. This trial will therefore investigate the effectiveness of a nurse-led educational intervention for adherence to DAAs in a PWID population.

Whilst the combination of Grazoprevir and Elbasvir is licensed for treatment of HCV genotype 1, treatment of HCV genotype 3 is more problematic. The C-SWIFT trial has recently shown that the combination of Grazoprevir, Elbasvir and Sofosbuvir is an effective and safe 8 week treatment for HCV genotype 3, resulting in high SVR rates. Whilst all 3 drugs are licensed for treatment of HCV, the combination is not yet licensed. This combination will be used to treat HCV genotype 3 infections in this trial.

Hepatitis C virus is prone to develop resistance to DAAs since it has a high replication rate and therefore forms large numbers of genetically-distinct viral variants. The investigators will investigate whether participants who do not achieve SVR are infected with a drug resistant strain of HCV by sequencing the NS3 and NS5A regions of viral nonstructural (NS) protein present within their blood. The proteins of these genes are targeted by the DAA medications and if their structure is altered the DAA may no longer be effective.

The trial will also explore whether the taking of illicit drugs affects the efficacy of treatment. While the main effect is likely to be via adherence, it is also possible that some of the illicit drugs may interact with the DAAs. A log of illicit drugs used by the participants will be kept and used to identify any candidate interactions for further investigation.

This is a randomised, un-blinded trial which will be conducted in the needle exchange services and pharmacies across Tayside, designed to evaluate the efficacy and feasibility of DAA therapy, in HCV positive, genotype 1 and 3, active PWIDs, administered via three different routes:

1. DOT,
2. Fortnightly pick-up
3. Fortnightly pick-up with psychological intervention.

Participants included in the trial will have a reactive Dry Blood Spot (DBS) test to confirm HCV infection, polymerase chain reaction (PCR) test to confirm active infection and will currently be using illicit drugs, as confirmed by the participant. Drug screening (by urine sample) will not be tested at that time.

Participants will be stratified by the genotype of their HCV infection; genotype 1 vs genotype 3 and randomised to one of three groups; DOT, fortnightly pick-up, or fortnightly pick-up with psychological adherence intervention.

All PWID are encouraged to have a DBS test annually as part of clinical practice in Tayside. Upon receipt of a reactive DBS test, potential participants will be briefed about the trial by the specialist nurse or other trained member of staff and given a participant information sheet (PIS) informing them of what is involved. Willing individuals will provide written informed consent and will then have safety bloods drawn to determine eligibility to proceed.

Participants in all three arms of the trial will attend a baseline visit, a randomisation visit either one (genotype 3) or two (genotype 1) visits during treatment, an end of treatment visit and an SVR visit.

All participants will be given incentives to continue with their treatment in the trial. These will consist of protein drinks and will be given at each study visit.

Psychological intervention Participants randomised to fortnightly pick-up with psychological intervention will have an interview with the study nurse, prior to beginning their treatment, which will cover the educational intervention designed to aid their compliance with the drug regimen. The intervention will be based on the Information-Motivation-Behavioural (IMB) Skills Model of Adherence12 which was originally developed to explain adherence behaviour in HIV. Recent research suggests this model may have applicability in understanding the facilitator and barriers to adherence in HCV patients. The model suggests that provision of medication information, enhancing personal and social motivation and developing behavioural skills that are key determinants of adherence and may improve adherence in this group. The intervention will involve a structured interview in which the trial nurse and participant will develop an action plan that includes personalised information, sources of motivation for adherence and a treatment routine configured to be compatible with the participant's lifestyle. Anticipating barriers to adherence and problem-solving will be included in the treatment routine. The intervention will take place at the randomisation visit and last approximately one hour. During the intervention, participants will be guided by their trial nurse in the completion of a personalised booklet, "Hepatitis C and Me". The booklet contains general and personalised information on Hepatitis C, exercises designed to explore and enhance personal and social motivation for treatment adherence and a behavioural action plan (the skills element of the IMB model). The booklet uses the principles of node-link mapping to structure the intervention. Node link mapping use a set of visual tools to structure and guide therapeutic conversation and has been shown to enhance memory and compliance with treatment in substance misusers. Participants in the other two arms of the trial, who are not receiving the psychological intervention, will be given the current National Health Service (NHS) Tayside hepatitis information booklet ("Living with Hepatitis C") which provides generalised information about HCV without personalised information or specific strategies to enhance motivation and behavioural skills.

Reinfection follow up. Trial participants will be invited to also consent for access to information from their annual clinic visits and HCV testing at any other contact with clinical services for up to 5 years, to detect re-infection.

Illicit drug monitoring Illicit drug use will be recorded at baseline and at end of treatment (week 8 for genotype 3, week 12 for genotype 1). One sample of urine for toxicology will be taken during treatment. Those participants who fail to achieve SVR will be compared to successful participants for any correlation with particular substance use. For any candidate substance associated with failure to achieve SVR not explained by lack of adherence, biological samples will be analysed for biological mechanisms.

Adherence monitoring Adherence of those participants randomised to DOT will be documented on a daily log. Those randomised to fortnightly collection of medication will receive Zepatier tablets in blister packaging. They will return their packets of medication every two weeks and any remaining tablets will be counted. Participants infected with HCV genotype 3 will additionally receive bottles containing Sovaldi tablets. These bottles will be fitted with adherence aid caps that record time and date of each cap opening.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female. (Age limit 18-70)
* HCV PCR confirmed active infection, genotype 1 or 3.
* If female, must have negative urine test results for pregnancy during initial screening period (for trial inclusion) and be advised of limited safety data in pregnancy.
* Current illicit drug use established through participant history.
* Able to provide informed consent, agreeing to trial and clinical monitoring criteria

Exclusion Criteria:

* Aggressive or violent behaviour.
* Platelet count < 75000000000 /ml
* Alanine transaminase > 350 Units/l
* Inability to provide informed consent.
* Clinical history or abnormal valves for albumin< 30 g/l, Bilirubin >35 umol/l or prothrombin time >1.5 consistent with decompensated liver failure Childs-Pugh B or C
* Clinical history of primary hepatocellular carcinoma
* Pregnancy or breast feeding.
* Participation in a drug trial within the previous 30 days
* Hepatitis B surface antigen positive
* HIV infection.
* Hypersensitivity to elbasvir and grazoprevir
* Hypersensitivity to sofosbuvir (genotype 3 infected-participants ony)
* Currently being treated with an inhibitor of organic anion transporting polypeptide 1B, e.g. rifampicin, atazanavir, daruavir, lopinavir, saquinavir, tipranavir, cobicistat or ciclosporin.
* Currently being treated with inducers of cytochrome P450 3A or P-glycoprotein, such as efavirenz, phenytoin, carbamazepine, bosentan, etravirine, modafinil or St John's Wort (Hypericum perforatum)
* Currently being treated with amiodarone (Participants infected with genotype 3 HCV only)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Dillon, MD, Principal Investigator — University of Dundee
Locations (2):
- United Kingdom (2):
  - University of Dundee, Dundee, Tayside
  - NHS Tayside, Dundee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beer L, Inglis S, Malaguti A, Byrne C, Sharkey C, Robinson E, Gillings K, Radley A, Hapca A, Stephens B, Dillon J. Randomized clinical trial: Direct-acting antivirals as treatment for hepatitis C in people who inject drugs: Delivered in needle and syringe programs via directly observed therapy versus fortnightly collection. J Viral Hepat. 2022 Aug;29(8):646-653. doi: 10.1111/jvh.13701. Epub 2022 May 26. PMID 35582875
- [Derived] Inglis SK, Beer LJ, Byrne C, Malaguti A, Robinson E, Sharkey C, Gillings K, Stephens B, Dillon JF. Randomised controlled trial conducted in injecting equipment provision sites to compare the effectiveness of different hepatitis C treatment regimens in people who inject drugs: A Direct obserVed therApy versus fortNightly CollEction study for HCV treatment-ADVANCE HCV protocol study. BMJ Open. 2019 Aug 8;9(8):e029516. doi: 10.1136/bmjopen-2019-029516. PMID 31399460

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 135 participants were recruited. 6 withdrew by choice prior to randomisation. One randomised participant had to be withdrawn prior to starting treatment due to elevated Alanine Aminotransferase (ALT) levels, over the limit for inclusion in this study. Hence 128 participants who initiated treatment.
Groups:
- Daily Observed Therapy: Patients with active hepatitis C infection genotype 1 will receive 12 weeks treatment with Zepatier at one tablet per day. Patients with active hepatitis C infection genotype 3 will receive 8 weeks treatment with Zepatier pill plus Sofosbuvir pill at one of each tablets per day. These tablets will be given to patients on a daily, observed basis by either the nurse or a community pharmacist.
  Zepatier Pill: Drugs will be given to participants to treat hepatitis C infection
  Sofosbuvir Pill: Drugs will be given along with Zepatier to participants to treat genotype 3hepatitis C infection
- Fortnightly Pick-up: Patients with active hepatitis C infection genotype 1 will receive 12 weeks treatment with Zepatier at one tablet per day. Patients with active hepatitis C infection genotype 3 will receive 8 weeks treatment with Zepatier pill plus Sofosbuvir pill at one of each tablets per day. These tablets will be given to patients on a fortnightly basis by the nurse.
  Zepatier Pill: Drugs will be given to participants to treat hepatitis C infection
  Sofosbuvir Pill: Drugs will be given along with Zepatier to participants to treat genotype 3hepatitis C infection
- Fortnightly Pick-up +Psych Intervention: Patients with active hepatitis C infection genotype 1 will receive 12 weeks treatment with Zepatier at one tablet per day. Patients with active hepatitis C infection genotype 3 will receive 8 weeks treatment with Zepatier pill plus Sofosbuvir pill at one of each tablets per day. These tablets will be given to patients on a fortnightly basis by the nurse. In addition, this group will receive a one-off interview with the researcher to complete a psychological intervention designed to improve adherence to the medication regimen.
  Zepatier Pill: Drugs will be given to participants to treat hepatitis C infection
  Psychological intervention: Participants randomised to fortnightly pick-up with psychological intervention will have an interview with the study nurse designed to aid their compliance with the drug regimen. During the intervention participants will be guided by their trial nurse in the completion of a personalised booklet, "Hepatitis C and Me". The booklet uses the principles of node-link mapping to structure the intervention.
  Sofosbuvir Pill: Drugs will be given along with Zepatier to participants to treat genotype 3hepatitis C infection
Period: Overall Study
Arm/Group | Daily Observed Therapy | Fortnightly Pick-up | Fortnightly Pick-up +Psych Intervention
Started | 39 | 42 | 47
Completed | 33 | 37 | 40
Not Completed | 6 | 5 | 7
Not completed — Death | 1 | 1 | 1
Not completed — Withdrawal by Subject | 3 | 3 | 4
Not completed — Did not initiate treatment | 2 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Daily Observed Therapy | Fortnightly Pick-up | Fortnightly Pick-up +Psych Intervention | Total
Number analyzed (Participants) | 39 | 42 | 47 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (8.20) | 35.7 (7.33) | 37.7 (7.53) | 36.6 (7.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 15 | 36
  Male | 29 | 31 | 32 | 92
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 39 | 42 | 47 | 128
Living Situation [Count of Participants; unit: Participants] — Type of living accommodation used by participants
  Participants
    Owned/rented | 24 | 24 | 31 | 79
    Supported accommodation (drug related) | 1 | 3 | 2 | 6
    Homeless | 13 | 13 | 12 | 38
    Other | 1 | 2 | 2 | 5
Source of income [Count of Participants; unit: Participants]
  Unemployed on government benefit | 20 | 23 | 30 | 73
  Unemployed on government benefit and at least one other source of income | 18 | 15 | 14 | 47
  Casual work and government benefit | 1 | 1 | 0 | 2
  No government benefit but other source of income | 0 | 3 | 3 | 6
Alcohol consumption [Count of Participants; unit: Participants]
  None | 32 | 33 | 37 | 102
  Between 1-20 units | 5 | 8 | 8 | 21
  Over 20 units | 2 | 1 | 2 | 5
Drug injecting history [Count of Participants; unit: Participants]
  Injected within last week | 27 | 28 | 33 | 88
  Injected within last month | 4 | 8 | 6 | 18
  Injected within last 3 months | 8 | 6 | 8 | 22

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Sustained Viral Response at 12 Weeks Post Treatment (SVR12) in the Three Treatment Groups.
Description: SVR12 of participants in the directly observed therapy (DOT), fortnightly pick-up or fortnightly pick-up with a psychological adherence intervention group. SVR12 was measured by viral load of hepatitis c virus (HCV) in participant's blood at least 12 weeks after end of treatment. A viral load of less than 10IU/ml indicates no active infection and SVR12 has been achieved.
Time Frame: 24 weeks for genotype 1 HCV, 20 weeks for genotype 3 HCV infection
Measure: Count of Participants; unit: Participants
Arm/Group | Daily Observed Therapy | Fortnightly Pick-up | Fortnightly Pick-up +Psych Intervention
Number analyzed (Participants) | 33 | 37 | 40
Participants
  SVR test positive for virus | 3 | 5 | 3
  SVR test negative for virus | 30 | 32 | 37
Statistical Analysis 1: Comparison: Daily Observed Therapy vs Fortnightly Pick-up; Test type: Non-Inferiority — Assuming a 95% SVR rate (based on published studies) in the DOT arm of the trial in this population and a non-inferiority limit of 14% (which would be likely to maintain cost-effectiveness) then at a 5% significance level and 90% power we would need a sample size of 42 in each group 126 in total. To allow for drop-outs we will aim to recruit 135 individuals, 45 per group; p = 0.67, Logistic; Odds Ratio (OR) = 0.64, 95% CI 2-sided [0.14 to 3.00]
Statistical Analysis 2: Comparison: Fortnightly Pick-up vs Fortnightly Pick-up +Psych Intervention; Test type: Non-Inferiority — Described in Statistical Analysis 1; p = 0.41, logistic; Odds Ratio (OR) = 0.53, 95% CI 2-sided [0.11 to 2.45]
Statistical Analysis 3: Comparison: Daily Observed Therapy vs Fortnightly Pick-up +Psych Intervention; Test type: Non-Inferiority — Described in Statistical Analysis 1; p = 0.82, logistic; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.23 to 6.61]

2. Secondary Outcome: Adherence as Assessed by the Total Percentage of Tablets Taken (Out of Those Dispensed) During the Treatment Period
Description: Adherence of daily directly observed therapy group from daily logs Adherence measured by counting tablets returned after each 2 week treatment period (fortnightly pickup groups) Adherence of participants infected with genotype 3 and treated with Sovaldi measured using medication event monitoring system (MEMS®) cap.
Time Frame: 12 weeks for genotype 1 HCV, 8 weeks for genotype 3 HCV infection
Measure: Mean (Standard Deviation); unit: percentage of medication taken
Arm/Group | Daily Observed Therapy | Fortnightly Pick-up | Fortnightly Pick-up +Psych Intervention
Number analyzed (Participants) | 39 | 42 | 47
percentage of medication taken | 69 (0.32) | 96 (0.09) | 98 (0.05)

3. Secondary Outcome: Assessment of Reinfection Rates in Active PWIDs Treated With Oral DAA Regimes
Description: Hepatitis C viral load by polymerase chain reaction (PCR) analysis. Any participants testing positive for reinfection post SVR12.
  This data will no longer be collected as part of this study and will be collected as part of standard clinical care.
Time Frame: Not applicable. Not part of study data set.
Population: Data not collected.
Arm/Group | Daily Observed Therapy | Fortnightly Pick-up | Fortnightly Pick-up +Psych Intervention
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Assessment of Resistance Profiles in Those Who do Not Achieve SVR
Description: Profiles of the HCV viral resistance proteins, NS5a and NS3 in participants who did not achieve SVR12, for reasons other than non-adherence to treatment.
Time Frame: Bloods collected at baseline, end of treatment and 12 weeks post end of treatment
Population: Viral resistance would be tested for in instances where a positive HCV blood test at the SVR12 stage could not be explained by non-adherence to medication. No participants met this criteria.
Arm/Group | Daily Observed Therapy | Fortnightly Pick-up | Fortnightly Pick-up +Psych Intervention
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Assessment of the Types of Illicit Drugs Taken by Trial Participants and Identification of Any Interaction With the Directly Acting Therapies.
Description: Drug misuse history and urine toxicology to test for potential illicit drug interactions with the treatment in participants who did not achieve SVR12 for reasons that are not non-adherence to treatment.
Time Frame: At three timepoints; time zero (before treatment), time 2-8 weeks (during treatment) time 12 weeks (at the end of treatment)
Population: Toxicological analysis of participant's urine for potential interacting illicit drugs would be tested for in instances where a positive HCV blood test at the SVR12 stage could not be explained by non-adherence to medication. No participants met this criteria.
Arm/Group | Daily Observed Therapy | Fortnightly Pick-up | Fortnightly Pick-up +Psych Intervention
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 31 months
Description: Recorded but not reported as Serious Adverse Events:
  * Death or hospitalisation for assault or accidental injury
  * Hospitalisation for abscesses due to drugs use
  * Hospitalisation for wound management due to drugs use
  * Death or hospitalisation due to infection
  * Hospitalisation for elective or planned investigation or treatment
  * Death or hospitalisation for deteriorating renal function, high or low potassium levels
  * Hospitalisation due to nausea, vomiting, constipation or diarrhea
Arm/Group | Daily Observed Therapy | Fortnightly Pick-up | Fortnightly Pick-up +Psych Intervention
All-Cause Mortality (participants affected / at risk) | 1/39 | 1/42 | 1/47
Serious Adverse Events (participants affected / at risk) | 6/39 | 9/42 | 8/47
Other Adverse Events (participants affected / at risk) | 8/39 | 10/42 | 6/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daily Observed Therapy (N=39) | Fortnightly Pick-up (N=42) | Fortnightly Pick-up +Psych Intervention (N=47)
Intentional self harm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Left mild cerebral infarct (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Mania (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 2 (3)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vascular psuedoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 2 (2) | 1 (1)
Illicit drug overdose (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Groin abcess (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Intervertebral discitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Community acquired pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Neck pain secondary to fall (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Loss of consciousness due to drug use (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Septic emboli (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Physical assault (Social circumstances) | 1 (1) | 0 (0) | 0 (0)
Streptococcus bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daily Observed Therapy (N=39) | Fortnightly Pick-up (N=42) | Fortnightly Pick-up +Psych Intervention (N=47)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 4 (4) | 1 (1)
Injection site infection/abscess (Infections and infestations) | 2 (2) | 3 (4) | 3 (9) — Infection or abscess related to injecting drug use
Illicit drug overdose (Injury, poisoning and procedural complications) | 5 (5) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-04-02): https://cdn.clinicaltrials.gov/large-docs/06/NCT03236506/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-29): https://cdn.clinicaltrials.gov/large-docs/06/NCT03236506/SAP_002.pdf